CLINICAL TRIAL: NCT05319145
Title: PeRsonalizing the Approach to the Oncologic Frail Individual Through Tailored Assessment and Intervention (PROFIT Study)
Acronym: PROFIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Servicio de Geriatría Complejo Hospitalario de Navarra (CHN) (Unknown); Fundación Miguel Servet - Navarrabiomed (Unknown); Hospital de la Ribera, Alzira, Valencia (Unknown); Institut Català d'Oncologia ICO Girona (Unknown); Vall d'Hebron Institute of Oncology (Other); Servei Andorrà d'Atenció Sanitària (SAAS), Andorra (Unknown); Gemelli Hospital, Universidad Cattolica del Sacro Cuore, Roma (Italia) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROFIT Study
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Older Adults; Gastro-Intestinal Cancer; Prostate Cancer; Lung Cancer; Frail Elderly Syndrome
MeSH Terms: conditions — Prostatic Neoplasms; Lung Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Treatment as usual. Mainly based on standard physical rehabilitation.
  Interventions: Other: Control group
- Intervention group (Experimental): Based on the results of the CGA, a tailored multidisciplinary intervention will be proposed, focused on a multicomponent physical exercise program with nutritional recommendations.
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — 1) Multi-component exercise intervention program based on Vivifrail©. It consists of 1 daily-30 minutes session, twice a week, for 10 consecutive weeks supervised by an experienced exercise specialist. Exercises (resistance, gait retraining, balance training) are personalized depending on the person's functional capacity (evaluated by the SPPB and a walking speed test) and the risk of falling. Between sessions, individual, unsupervised training by the own patient, supported in the case by the caregiver, will be stimulated, through the recommendations of ViviFrail©. 2) Nutrition. Personalized recommendations according to nutritional and medical status (active oncologic treatment, remission, or palliative stage) will be offered according to the ESPEN recommendations for cancer patients, aimed at compensating for inadequate energy intake, improving patients' malnutrition risk stage (assessed by means of the MNA-SF).
  Other Names: Tailored multidisciplinary intervention based on CGA, focused on a multicomponent physical exercise program with nutritional recommendations.
  Arms: Intervention group
Other: Control group — General recommendations (written and videos) will be offered.
  Other Names: Health psycho-education
  Arms: Control group

SUMMARY:
The PROFIT study has two complementary aims. The first aim is to compare, in a cohort study enrolling N=257 older adults (>65 years) with lung, gastrointestinal and prostate cancer, different easy measures of frailty (Geriatric 8 questionnaire (G8), Short physical Performance Battery (SPPB) and the IF-VIG), testing their ability to predict survival, functional status (ECOG, Barthel Index), quality of life (EuroQol5D) and resources utilization (visits, hospital admissions, treatments) at 3, 6 and 12 months. The second aim, which motivates the registration in ClinicalTrials.gov, is to conduct a randomized controlled trial (RCT) enrolling N=134 patients per group, with similar characteristics to those enrolled for aim 1, but with mild-moderate frailty (G8≤14 points); we will compare a multi-component CGA-based intervention including physical exercise and nutritional recommendations with usual care, measuring the impact on the same outcomes as for aim 1, at 3 and 6 months. The use of ad hoc eHealth solutions (App/platform for exercise) will foster patients' empowerment and sustainability of the intervention. We will also assess patients, caregivers, and professionals' experience with the intervention through focus groups. Participants will be recruited from outpatients and from post-acute care units.

DETAILED DESCRIPTION:
The impact of the aging of population on cancer incidence and consequences is clear: in very few years, more than 50% of older adults will be diagnosed with malignant tumors, with a relevant increase in mortality compared to younger adults, and a dramatic burden of disability. Many of these patients will be potential candidates for oncospecific treatments, either curative, adjuvants or palliative. Despite this scenario, many trials on cancers still exclude patients based on their age or set survival and treatments' toxicity as the main outcomes, neglecting other meaningful outcomes such as functional status or quality of life. Therefore, clinical decisions regarding this specific population are not always based on real-life data. Moreover, older adults are a highly heterogeneous population, based on clinical, functional, and psychosocial aspects. This is why, in such a population group, the individualization of treatments is pivotal.

Frailty has been proposed as a better marker of biological age than chronological age. This concept indicates a reversible state of risk of increased vulnerability to external or internal stressors, exposing the patients to a higher risk of adverse events, including disability and mortality. However, there is no agreement on the most suitable frailty tools to be used in practice. In older adults with cancer, frailty, which is easily measured in any setting through quick clinical scales, could be an ideal trigger to select candidate patients for a subsequent more extensive comprehensive geriatric assessment (onwards, CGA) and potential interventions. Among these interventions, multi-component approaches including physical exercise and nutritional recommendations have shown a positive impact on both mortality and functional status in patients with different cancers and could be proposed for either pre-habilitation or re-habilitation in older cancer patients with mild-moderate frailty.

Considering these premises, the PROFIT study has two complementary aims. The first aim is to compare, in a cohort study enrolling N=257 older adults (>65 years) with lung, gastrointestinal and prostate cancer, different easy measures of frailty (Geriatric 8 questionnaire (G8), Short physical Performance Battery (SPPB) and the IF-VIG), testing their ability to predict survival, functional status (ECOG, Barthel Index), quality of life (EuroQol5D) and resources utilization (visits, hospital admissions, treatments) at 3, 6 and 12 months. The second aim is to conduct a randomized controlled trial (RCT) enrolling N=134 patients per group, with similar characteristics to those enrolled for aim 1, but with mild-moderate frailty (G8≤14 points); we will compare a multi-component CGA-based intervention including physical exercise and nutritional recommendations with usual care, measuring the impact on the same outcomes as for aim 1, at 3 and 6 months. The use of ad hoc eHealth solutions (App/platform for exercise) will foster patients' empowerment and sustainability of the intervention. We will also assess patients, caregivers, and professionals' experience with the intervention through focus groups. Participants will be recruited from outpatients and from post-acute care units.

The PROFIT study will add relevant evidence for the management of older cancer patients. The impact, for the individual and the society, is high, in light of the aging of the population: the results will allow providing oncologists and other professionals with tools to improve the personalization of treatments, to finally provide adequate and tailored care programs. This might contribute to avoid the exclusion of patients who could benefit from active treatments and, on the other hand, reducing overtreatment for those who will likely not benefit from it. The clinical trial will also provide information on the most suitable content and on the impact of an intervention aimed at strengthening the functional status and improving the quality of life in older cancer patients with mild-moderate frailty, who might be potential candidates for subsequent onco-specific treatments. The project will also deliver adapted materials and eHealth solutions to be potentially scaled up for this profile of users, as a benefit for the society even beyond this project.

ELIGIBILITY:
Inclusion Criteria:

1) Older adults (≥65 years) 2) Diagnosed with solid tumors (specifically, prostate, lung, colon, rectal, hepatic-biliary, pancreatic, and esophagus-gastric cancers), an extension of T2, T3, T4, involving or not lymph nodes, and either metastatic or not (M0-1), who might or might not underwent onco-specific treatments or await for new treatments 3) Evidence of functional impact (ECOG≥2) but overall maintained functional status (Barthel≥50) 4) Life expectancy ≥3 months 5) Patients with mild-moderate frailty (G8<14) 5) Willing to provide informed consent to participate.

Exclusion Criteria:

1) Participants with moderate-severe cognitive impairment (Reisberg's Global Deterioration Scale ≥5).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Change in physical function, measured by the difference on SPPB between follow-ups, hand grip and maximum resistance.

SECONDARY OUTCOMES:
Barthel | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Functional status and disability
ECOG | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Functional status and disability
EQoL-5D | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Quality of life
Edmonton Symptom Assessment System | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Intensity of specific symptoms related to cancer
Falls (yes vs. no & number of events) | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Potential adverse effects of the intervention
Fractures (yes vs. no & number of events) | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Potential adverse effects of the intervention
Pain (0-10 VAS) | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Potential adverse effects of the intervention
Cardiovascular events (yes vs. no & number of events) | Pre-intervention (baseline) and post-intervention at follow-ups (at 3, 6, and 12 months)
  Collecting ocurrence of angina, myocardial infarction, TIA and/or stroke
Readmissions to the acute hospital | Post-intervention at follow-ups (at 3, 6, and 12 months)
  Potential adverse effects
Days spent at home (number of days) | Post-intervention at follow-ups (at 3, 6, and 12 months)
  Related to process & resources utilization

CONTACTS AND LOCATIONS:
Locations (3):
- Servei Andorrà d'Atenció Sanitària, Andorra la Vella, Andorra, Andorra
- Spain (2):
  - NavarraBiomed, Pamplona, Navarre
  - Parc Sanitari Pere Virgili - Vall d'Hebron Institut de Recerca, Barcelona